CLINICAL TRIAL: NCT07220226
Title: Venous Function and the Effect of Venous Compression on Exercise Cardiovascular Function in Patients With Fontan Circulation.
Brief Title: Venous Compression in Fontan
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Keri Shafer, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: STU20250885
Record Dates: First submitted 2025-09-25; First posted 2025-10-23 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-10

CONDITIONS: Single-ventricle; Fontan Circulation
Keywords: Venous Compression; Exercise Testing; Cardiac Reserve; Fontan Circulation; Magnetic Resonance Imaging; vascular function
MeSH Terms: conditions — Univentricular Heart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Fontan circulation Arm (Experimental): Fontan circulation participants will undergo Rest +Submax exercise with and without wearing venous compression garments.
  A subset of patients with Fontan circulation will undergo repeat testing 2-weeks later.
  Interventions: Device: Lower extremity compression garments; Other: Without compression garments
- Healthy controls (Experimental): Healthy group participants will undergo Rest +Submax exercise with and without wearing venous compression garments.
  Interventions: Device: Lower extremity compression garments; Other: Without compression garments

INTERVENTIONS:
Device: Lower extremity compression garments — Acute and 2-week effects of compression garments
Other: Without compression garments — Acute effects without compression garments

SUMMARY:
The aim of this study is to investigate whether venous compression garments increase exercise stroke volume in patients with Fontan circulation. To address this aim, we will test the following hypotheses:

1. Acute and chronic external venous compression will increase exercise stroke volume in patients with Fontan circulation.
2. Patients with significant venous varicosities will have a greater response to venous compression.

Participants will:

* Undergo submaximal exercise testing in MRI to measure venous return and exercise stroke volume with and without the wearing of compression garments
* Undergo submaximal exercise testing on a seated upright exercise ergometer with concurrent measurement of stroke volume with and without the wearing of compression garments
* A subset of participants will repeat both testing visits after wearing compression garments for 2-weeks during waking hours.

Participants will:

* Undergo submaximal exercise testing in MRI to measure venous return and exercise stroke volume with and without the wearing of compression garments
* Undergo submaximal exercise testing on a seated upright exercise ergometer with concurrent measurement of stroke volume with and without the wearing of compression garments
* A subset of participants will repeat both testing visits after wearing compression garments for 2-weeks during waking hours.

DETAILED DESCRIPTION:
Study Day 1 - Consent, Screening and Garment Measurements:

Following assessment of participant eligibility, all participants will undergo leg venous ultrasound assessment and abdominal-foot measurements for the custom making of compression garments.

Study Day 2 - MRI:

Study participants will undergo comprehensive cardiovascular MRI using a 3T MRI scanner with and without compression garments and exercise.

Study Day 3 - Cardiovascular & Exercise Testing Day:

All participants will undergo comprehensive cardiovascular structure and function assessments at rest and during exercise with and without the wearing of compression garments. Baseline testing will include dual x-ray absorptiometry (DEXA), pulmonary function testing, comprensive vascular assessments and echocardiography. During exercise at two submaximal workloads, the study team will measure blood pressure, oxygen uptake and cardiac output.

ELIGIBILITY:
Patients with a Fontan circulation -

Inclusion criteria:

• Patients at UTSW aged 18-45 years old with a Fontan circulation.

Exclusion Criteria:

* NYHA Class 4
* Severe AV valve regurgitation
* Severe ventricular dysfunction
* Large ascites
* Significant varicosities
* Atrio-pulmonary (AP) Fontan
* Known Fontan thrombus
* Poorly controlled arrythmia
* Unplanned cardiac admission in the last 6 months
* Cyanosis (resting O2 saturation <85%)
* Pregnant
* Common femoral vein obstruction >50% to be performed following completion of informed consent.

Healthy Controls:

Healthy control participants will be recruited on the basis of having no known chronic diseases and not currently taking any cardiovascular medications.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Stroke Volume with Exercise | Rest (20 minutes), Exercise (10 minutes)
  The change in single ventricular stroke volume from rest to moderate intensity exercise with compression garments during baseline testing
Change in Stroke Volume with Exercise | Rest (20 minutes), Exercise (10 minutes)
  The change in single ventricular stroke volume from rest to moderate intensity exercise without compression garments during baseline testing
Change in Stroke Volume with Exercise | Rest (20 minutes), Exercise (10 minutes) at 2-weeks follow-up testing
  The change in single ventricular stroke volume from rest to moderate intensity exercise following 2 weeks of wearing compression garments.
The Acute Effect of Compression Garments on Stroke Volume during Exercise | Rest (20 minutes) and Exercise (10 minutes) repeated during baseline testing
  The difference in the change in single ventricular stroke volume during moderate intensity exercise between baseline testing with (outcome #1) and without (outcome #2) garments
The Chronic Effect of Compression Garments on Stroke Volume during exercise | Rest (20 minutes) and Exercise (10 minutes) completed during baseline and during follow-up testing
  The difference in the change in single ventricular stroke volume during moderate intensity exercise between baseline testing without garments (outcome #2) and following 2 weeks of wearing compression garments (outcome #3) in patients with Fontan Circulation.

SECONDARY OUTCOMES:
Change in Venous Return with Exercise | Rest (10 minutes) and Exercise (5 minutes)
  The change in inferior vena cava flow from rest to moderate intensity exercise with compression garments using MRI during baseline testing
Change in Venous Return with Exercise | Rest (10 minutes) and Exercise (5 minutes)
  The change in inferior vena cava flow from rest to moderate intensity exercise without compression garments using MRI during baseline testing
Change in Venous Return with Exercise | Rest (10 minutes) and Exercise (5 minutes)
  The change in inferior vena cava flow from rest to moderate intensity exercise following 2 weeks of wearing compression garments using MRI
The Acute Effect of Compression Garments on Changes in Venous Return with Exercise | Rest (10 minutes) and Exercise (5 minutes) repeated during baseline testing
  The difference in the change in inferior vena cava flow during moderate intensity exercise between baseline testing with (outcome #6) and without (outcome #7) garments
The Chronic Effect of Compression Garments on Changes in Venous Return with Exercise | Rest (10 minutes) and Exercise (5 minutes) completed during baseline and during follow-up testing
  The difference in the change in inferior vena cava flow during moderate intensity exercise between baseline testing without garments (outcome #7) and following 2 weeks of wearing compression garments (outcome #8) in patients with Fontan Circulation.

CONTACTS AND LOCATIONS:
Overall Officials: Keri Shafer, MD, Principal Investigator — University of Texas Southwestern Medical Center

IPD SHARING:
Plan to Share IPD: No